CLINICAL TRIAL: NCT04276090
Title: Feasibility Pilot of Hepatic Arterial Infusion Chemotherapy in a Rural Catchment Area, Using the Codman Vascular Catheter With the Synchromed II Pump, for Patients With Unresectable Colorectal Cancer Liver Metastases or Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Codman Catheter/Synchromed Pump Hepatic Artery Chemotherapy for Unresectable Colorectal Metastases/Intrahepatic Cholangiocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: an alternate device became FDA approved
Sponsor: Michael J Cavnar, MD (Other)
Responsible Party: Sponsor-Investigator, Michael J Cavnar, MD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19-GI-109-PMC
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Bile Duct Neoplasms; Colorectal Neoplasms
Keywords: hepatic artery infusion pump; colorectal liver metastases; intrahepatic cholangiocarcinoma; FUDR; floxuridine
MeSH Terms: conditions — Bile Duct Neoplasms; Colorectal Neoplasms; Cholangiocarcinoma | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients with unresectable colorectal liver metastases (arm 1) and unresectable intrahepatic cholangiocarcinoma (arm 2), will undergo hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter. All patients will receive hepatic artery infusion floxuridine, and then individual arms will receive disease-specific systemic chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Colorectal liver metastases (Experimental): Patients with unresectable colorectal liver metastases will undergo hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter. Patients will then receive hepatic artery infusion floxuridine as well as disease-appropriate systemic chemotherapy (FOLFOX, FOLRIRI, or oxaliplatin/irinotecan, or panitumumab if KRAS/NRAS wild type)
  Interventions: Device: Hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter.; Drug: Hepatic artery infusion pump floxuridine and dexamethasone; Drug: Systemic chemotherapy for colorectal liver metastases
- Intrahepatic cholangiocarcinoma (Experimental): Patients with unresectable intrahepatic cholangiocarcinoma will undergo hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter. Patients will then receive hepatic artery infusion floxuridine as well as disease-appropriate systemic chemotherapy (gemcitabine/oxaliplatin or gemcitabine alone)
  Interventions: Device: Hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter.; Drug: Hepatic artery infusion pump floxuridine and dexamethasone; Drug: Systemic chemotherapy for intrahepatic cholangiocarcinoma

INTERVENTIONS:
Device: Hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter. — Patients will undergo surgical hepatic artery infusion pump placement using the Synchromed II pump and the Codman tapered arterial catheter.
Drug: Hepatic artery infusion pump floxuridine and dexamethasone — Patients will receive infusion of floxuridine (FUDR) and dexamethasone via hepatic artery infusion through the implanted pump
Drug: Systemic chemotherapy for colorectal liver metastases — Patients will receive disease-appropriate systemic chemotherapy for colorectal liver metastases (FOLFOX, FOLFIRI, or irinotecan/oxaliplatin, or panitumumab if KRAS/NRAS wild type)
  Arms: Colorectal liver metastases
Drug: Systemic chemotherapy for intrahepatic cholangiocarcinoma — Patients will receive disease-appropriate systemic chemotherapy for intrahepatic cholangiocarcinoma (gemcitabine/oxaliplatin or gemcitabine alone)
  Arms: Intrahepatic cholangiocarcinoma

SUMMARY:
Due to discontinuation of the Codman C3000 pump, an alternate device is necessary to continue serving patients in need of hepatic arterial infusion chemotherapy. This study aims to test the safety of hepatic artery infusion pump placement, a standard surgical procedure, and intraarterial chemotherapy initiation with the standard medication floxuridine (FUDR), using the Medtronic Synchromed II pump combined with the Codman arterial catheter in patients with unresectable (not removable by surgery) liver metastases from colorectal cancer and unresectable intrahepatic cholangiocarcinoma. This study will determine if complication and pump loss rates will be similar to previously published rates for the Codman system.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Histologically confirmed unresectable colorectal adenocarcinoma metastatic to the liver with no definitive clinical or radiographic evidence of extrahepatic disease. Clinical or radiographic evidence of metastatic disease to peri-hepatic lymph nodes will be allowed, provided it is amenable to resection.

(OR)

* Histologically confirmed unresectable non-metastatic intrahepatic cholangiocarcinoma, with presence of less than 70% liver involvement. Clinical or radiographic evidence of metastatic disease to peri-hepatic lymph nodes will be allowed, provided it is amenable to resection.
* ECOG Performance Status of 0 - 1
* Lab Values ≤ 14 days prior to study enrollment:

absolute neutrophil count ≥1,500/mcL AST/ALT < 2.5 x institutional upper limit of normal (ULN) Platelets ≥ 100,000/mcL Creatinine < 1.5 mg/dL HGB > 9 g/dL Total Bilirubin ≤ 1.5 mg/dL

* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Prior chemotherapy is acceptable if last dose given ≥ 3 weeks prior to study enrollment.
* Any investigational agent is acceptable if last dose administered ≥ 3 months before study enrollment.

Exclusion Criteria:

* Presence of distant metastatic disease confirmed by radiographic evaluation. Clinical or radiographic evidence of metastatic disease to regional peri-hepatic lymph nodes will be allowed, provided it is amenable to resection.
* Prior radiation to the liver, including external beam, SBRT, Y90. Prior radiation therapy to the pelvis is acceptable.
* Active infection, hepatic encephalopathy
* Clinical evidence of portal hypertension (ascites, gastroesophageal varices or portal vein thrombosis; surgically-related ascites does not exclude the patient)
* Female patients who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female patients of child-bearing potential must have negative pregnancy test ≤72 hours before surgery)
* If in the opinion of the treating investigator a patient has any serious medical problems which may preclude receiving this type of treatment
* Patients with history or known presence of primary CNS tumors, seizures not well-controlled with standard medical therapy, or history of stroke
* Serious or non-healing active wound, ulcer, or bone fracture
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the HAIP chemotherapy (i.e., investigational regimen)
* Patients with psychiatric illness or social situations that would limit compliance with study requirements. Examples include: active substance abuse, active severe EtOH abuse, etc.
* Inability to reliably commit to traveling to Lexington, KY every 2 weeks for duration of the study treatment (6 months). Patient must have readily identifiable, reliable primary and back-up modes of transportation regardless of weather.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cavnar, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald HG, Cassim EB, Harper MM, Burke EE, Marcinkowski EF, Cavnar MJ, Pandalai PK, Kim J. The Development of Investigator-Initiated Clinical Trials in Surgical Oncology. Surg Oncol Clin N Am. 2023 Jan;32(1):13-25. doi: 10.1016/j.soc.2022.07.003. Epub 2022 Nov 3. PMID 36410913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Started | 17 | 4
Completed | 16 | 4
Not Completed | 1 | 0
Not completed — Rapid disease progression after surgery led to liver dysfunction; prevented administration of HAI | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma | Total
Number analyzed (Participants) | 17 | 4 | 21
Age, Customized [Count of Participants; unit: Participants]
  40-70 years | 17 | 4 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 4 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percent Completion of 1st Cycle of Hepatic Artery Chemotherapy
Description: The percent of patients who complete the 1st cycle of hepatic artery chemotherapy will be tabulated. This is a conglomerate safety endpoint which is a surrogate for any complication that prevents delivery of hepatic artery chemotherapy via the device combination.
Time Frame: approximately 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 16 | 4

2. Secondary Outcome: 30-day Postoperative Serious Adverse Events Related to Pump Implantation
Description: Tabulation of CTCAE serious adverse events attributed to pump implantation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 1 | 0

3. Secondary Outcome: 30-day Catheter Malfunction Due to Tubing Disconnect
Description: Quantify the percent of patients with inability to meet primary outcome due to catheter disconnects.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

4. Secondary Outcome: 30-day Catheter Malfunction Due to Inability to Access Pump
Description: Quantify the percent of patients with inability to meet primary outcome due to inability to access pump.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

5. Secondary Outcome: Percent of Patients That Require Secondary Intervention in Order to Obtain Primary Pump Function.
Description: Percentage of patients who need secondary intervention (IR embolization, revision of pump or tubing) to achieve primary pump function.
Time Frame: Approximately 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

6. Secondary Outcome: Percent of Screened Patients That Are Declined Due to High Risk of Failure as Determined by the Psychosocial Assessment Tool.
Description: Patients are screen using a psychosocial assessment tool for high risk of hepatic artery pump loss/failure, percent declined will be tabulated.
Time Frame: Immediate, determined at screening visit
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

7. Secondary Outcome: Percent Pump Loss Due to Inability to Attend Scheduled Followup Appointments.
Description: Percent of patients that experience pump loss/failure due to inability to attend scheduled followup appointments will be tabulated.
Time Frame: Approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

8. Secondary Outcome: Number of Interventions (Phone Calls) to Assure Patients Attend Followup Appointments.
Description: The number of staff contacts (phone calls) to assure patients keep their followup visits will be tabulated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 0 | 0

9. Secondary Outcome: Percent of Patients Who Remain on Hepatic Artery Infusion Pump Chemotherapy at 3 Months.
Description: The percentage of patients who remain on pump chemotherapy at 3 months will be tabulated.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 14 | 4

10. Secondary Outcome: Overall Response Rate at 6 Months
Description: RECIST v1.1 will be used to assess overall response rate at 6 months.
Time Frame: 6 months
Population: At the 6 month time point for this outcome there were only 14 evaluable participants for response rate due to attrition, death, or sub-RECIST threshold disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 11 | 3
Participants
  Progressive Disease | 4 | 2
  Stable Disease | 6 | 1
  Partial Response | 1 | 0

11. Secondary Outcome: Percent of Patients Who Are Downstaged and Undergo Surgery
Description: The percent of patients who are downstaged and undergo surgery will be tabulated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 7 | 0

12. Secondary Outcome: Percent of Patients Who Remain on Hepatic Artery Infusion Pump Chemotherapy at 6 Months.
Description: The percentage of patients who remain on pump chemotherapy at 6months will be tabulated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
Number analyzed (Participants) | 17 | 4
Participants | 13 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Colorectal Liver Metastases | Intrahepatic Cholangiocarcinoma
All-Cause Mortality (participants affected / at risk) | 3/17 | 2/4
Serious Adverse Events (participants affected / at risk) | 15/17 | 2/4
Other Adverse Events (participants affected / at risk) | 17/17 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Liver Metastases (N=17) | Intrahepatic Cholangiocarcinoma (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Other (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Immune system disorders) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Liver Metastases (N=17) | Intrahepatic Cholangiocarcinoma (N=4)
Anemia (Blood and lymphatic system disorders) | 15 (15) | 3 (3)
Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 6 (6) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 2 (2)
Other (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mucisitis Oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 12 (12) | 2 (2)
Fever (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (17) | 4 (4)
Alkaline phosphatase increased (Investigations) | 14 (14) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 17 (17) | 4 (4)
Blood bilirubin increased (Investigations) | 10 (10) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
INR increased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (11) | 3 (3)
Neutrophil count decreased (Investigations) | 7 (7) | 2 (2)
Platelet count decreased (Investigations) | 7 (7) | 4 (4)
White blood cell decreased (Investigations) | 5 (5) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (11) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Other (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (14) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 13 (13) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (12) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 10 (10) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT04276090/Prot_SAP_ICF_001.pdf